CLINICAL TRIAL: NCT03756441
Title: Effects of the Mindfulness-Based Health Promotion Program (MBHP) on the Quality of Life of Family Members of People With Intellectual Disability
Brief Title: Effects of the MBHP on the Quality of Life of Family Members of People With Intellectual Disability
Acronym: caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Mente Aberta de Mindfulness (Other)
Responsible Party: Principal Investigator, Marcelo Demarzo, MD, PhD, PhD, Centro Mente Aberta de Mindfulness
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 81973417.8.0000.5505
Record Dates: First submitted 2018-11-14; First posted 2018-11-28 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Quality of Life
MeSH Terms: interventions — Mindfulness; Psychotherapy, Group

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Mindfulness group (Experimental): This group will be included in the eight-week mindfulness program following the Mindfulness-Based Health Promotion protocol. They will group with have eight meetings, one per week, during a half hour and will learn the techiques to practice everyday during the week.
  Interventions: Behavioral: Mindfulness meditation
- Psychotherapy group (Active Comparator): This group will learn group problem solving techniques during eight weeks
  Interventions: Behavioral: Psychotherapy group

INTERVENTIONS:
Behavioral: Mindfulness meditation — This intervention is a meditative practice which the individuals will practive in their daily life following the MBHP protocol
  Arms: Experimental: Mindfulness group
Behavioral: Psychotherapy group — Caregivers will learn the technique of group problem solving
  Arms: Psychotherapy group

SUMMARY:
The research aims to verify the effects of the Mindfulness Based Health Promotion (PSBM) program on the quality of life of mothers of person with intellectual disability. Method: A randomized, controlled study with pre-post intervention measures and a follow-up measurement will be performed after six months of the end of the intervention. Sample: It will be composed of mothers of the 209 attended with moderate intellectual disability, adolescents and adults of the Service of Socioeducation of the Association of Parents and Friends of the Exceptional (APAE) of São Paulo, excluding those who have any psychiatric problem in the acute phase and minors, or who have regular practice of mindfulness or meditation in the last 6 months.

DETAILED DESCRIPTION:
Outcomes and Instruments to be used: As primary endpoint the quality of life of the family caregiver will be observed and as a secondary outcome the caregiver's overload will be observed. As explanatory variables will be considered anxiety, depression, functionality and level of attention to the present moment (mindfulness). The investigators will use focal group, Sociodemographic questionnaire, World Health Organization Disability Assessment Scale, Hospital Anxiety and Depression Scale, Brief Autocompaction Scale, World Health Organization Quality of Life Scale Brief Version, Mindful Attention Awareness Scale, Qualitative Analysis Questionnaire - Semi-Structured, Informal Caregiver Burden Assessment Questionnaire, Number of Practices and Adverse Effects. Procedure: The mothers of people with intellectual disability (ID) will be invited to participate in the research protocol. Having knowledge of the subject, agreeing to participate and signing the consent form, will respond to the questionnaires identified above, with a total duration of approximately 1 hour and 30 minutes. Subsequently the participants will be randomized into two groups, in which one will receive the mindfulness intervention and the other, active control, will participate in a Problem Solving Training. The protocols of questionnaires and focal group will be performed before, immediately after the accomplishment of the groups and in the follow-up of six months. The intervention group will last 8 weeks, according to the Mindfulness Based Health Promotion Program (PSBM) and during this same period the active control group will occur. Hypotheses and expected results: Mindfulness is expected to contribute to the improvement of the quality of life of this population, and so the investigators can contribute to the scientific increase in the theme.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years
* Being a mother with SASE DI
* Be in accordance with the Informed Consent Form

Exclusion Criteria:

* Under 18 years
* Acute psychiatric problem
* Regular practice of mindfulness or meditation in the last 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — In Brazil the number of female caregivers is higher than the male sex
Enrollment: 154 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of Life (WHOQOL-Bref) | 24 months
  Assess the impact of a Mindfulness-Based Health Promotion (MBHP) program on the quality of life by the WHOQOL-Bref of the family caregiver. Generic instrument of evaluation of the perception of the quality of life created by the World Health Organization (WHO). Abbreviated version, with 26 items grouped into 4 domains: physical, psychological, social and environmental health overall quality of life, and assessments by means of the average according to the quantity of issues in each domain. The results are presented according to the following score: 1-2,9 (good improvement), 3 -3,9 (regular), 4-4,9 (good), 5 (very good)

SECONDARY OUTCOMES:
Informal Caregiver Overload Assessment Questionnaire (QASCI) | 24 months
  Assess the Impact of a Mindfulness-Based Health Promotion Program on Overload of the caregiver. Questionnaire with 32 questions, developed in Portugal, adapted and validated for Brazil, was designed to measure the physical, emotional and social development of the informal caregiver with stroke, later used for informal caregivers of the elderly and dependent persons in at least one activity of daily living.
World Health Organization Disability Assessment Scale (WHODAS) | 24 months
  Assess the Impact of a Mindfulness-Based Health Promotion Program on Functionality of the caregiver. Designed to assess the level of functionality in six life domains (cognition, mobility, self-care, social coexistence, life activities and participation society), this scale covers the fields of International Classification of Functionality (CIF). The short version of 12 items will be used, translated and adapted to the Portuguese. The 'interviewer-administered' version will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo MP Demarzo, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Centro Mente Aberta de Mindfulness e Promoção de Saúde, São Paulo, São Paulo, Brazil